CLINICAL TRIAL: NCT01192412
Title: The CHIPS Trial (Control of Hypertension In Pregnancy Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Sunnybrook Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H08-00882; MCT-87522 (Other Grant/Funding Number: CIHR); 07-3431 (Other: UBC); NCT01081171 (obsolete NCT alias)
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Results first posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Gestational Hypertension
Keywords: hypertension; pregnancy; antihypertensive therapy; perinatal outcome; maternal outcome; Non-severe, non-proteinuric pre-existing or gestational hypertension in pregnancy
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 'Less tight' control. (Active Comparator): The diastolic blood pressure (dBP) treatment goal is 100 mmHg.
  Interventions: Procedure: Intervention is blood pressure management approach
- 'Tight' control. (Active Comparator): The diastolic blood pressure (dBP) treatment goal is 85 mmHg.
  Interventions: Procedure: Intervention is blood pressure management approach.

INTERVENTIONS:
Procedure: Intervention is blood pressure management approach — 1) 'Less tight' control. The dBP treatment goal is 100 mmHg. For safety, if dBP is >105 mmHg, then antihypertensive medication must be started or increased in dose. For dBP <100 mmHg, antihypertensive therapy should be decreased in dose or stopped, as appropriate. The intervention will be applied until delivery.
  Arms: 'Less tight' control.
Procedure: Intervention is blood pressure management approach. — 'Tight' control. The dBP treatment goal is 85 mmHg. For safety, if dBP is <80 mmHg, then antihypertensive medication must be decreased in dose or discontinued. If dBP is >85 mmHg, then antihypertensive therapy should be started or increased in dose. The intervention will be applied until delivery.
  Arms: 'Tight' control.

SUMMARY:
The investigators do not know which approach to treatment of non-severe high blood pressure in pregnancy is better for women and babies.

In the CHIPS Trial, the investigators seek to determine whether 'less tight' control (aiming for a diastolic blood pressure [dBP] of 100 mmHg), compared with 'tight' control (aiming for a diastolic blood pressure [dBP] of 85 mmHg) can decrease the risks of adverse baby outcomes without increasing the risk of problems for the mother.

DETAILED DESCRIPTION:
Primary research question:

For pregnant women with non-severe, non-proteinuric maternal hypertension at 14-33 weeks, will 'less tight' control (target diastolic blood pressure [dBP] of 100 mmHg) versus 'tight' control (target dBP of 85 mmHg) increase (or decrease) the likelihood of pregnancy loss or Neonatal Intensive Care Unit (NICU) admission for greater than 48 hours?

Secondary research question:

Will 'less tight' versus 'tight' control increase (or decrease) the likelihood of serious maternal complications?

Other research questions:

Will 'less tight' versus 'tight' control:

1. Increase (or decrease) the likelihood of serious perinatal complications?
2. Increase (or decrease) the likelihood of severe hypertension and pre-eclampsia?
3. Increase (or decrease) the likelihood of maternal satisfaction with care?
4. Result in significant changes in dBP or health care costs?

Treatment Allocation:

Eligible women will be randomised centrally to either 'less tight' control (aiming for dBP of 100mmHg) or 'tight' control (aiming for dBP of 85mmHg) of their hypertension.

Randomisation will be stratified by centre and type of hypertension (pre-existing or gestational).

* In the 'less tight' control group, if dBP is ≥105mmHg, then antihypertensive medication must be started or increased in dose.
* In the 'tight' control group, if dBP is ≤80mmHg, then antihypertensive medication must be decreased in dose or discontinued.
* In both groups, centres will provide their usual care. Data will be collected on potential co-interventions (e.g., hospitalisation, bedrest).

Outcomes:

Primary: Pregnancy loss (miscarriage or ectopic pregnancy, pregnancy termination, stillbirth, or neonatal death) or high level neonatal care for >48 hours in the first 28 days of life or prior to primary hospital discharge, whichever is later.

Secondary: One/more serious maternal complication(s) until six weeks postpartum.

Follow-up:

Compliance (dBP and antihypertensive dose) will be assessed within 4 weeks of randomisation. Outcome data will be collected during the woman's (and baby's) hospital stay for birth (or loss). Women will be contacted 6 to 12 weeks after delivery (or loss) and, for preterm babies, when the baby is at 36 weeks corrected gestational age to enquire about satisfaction with care and any major maternal/neonatal morbidity following hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-existing or gestational hypertension (pre-existing hypertension is dBP greater than or equal to 90 mmHg before pregnancy or 20 weeks' gestation; gestational hypertension is dBP greater than or equal to 90 mmHg that develops after 20 weeks)
2. dBP of 90 - 105 mmHg if NOT TAKING antihypertensive therapy, or dBP of 85 - 105 mmHg if TAKING antihypertensive therapy
3. Live foetus (confirmed by Doptone assessment of foetal heart tones within one week before randomisation)
4. Gestational age 14 - 33+6 weeks (as measured by last menstrual period or dating ultrasound)

Exclusion Criteria:

1. Severe systolic hypertension (defined as a systolic blood pressure [sBP] greater than or equal to 160 mmHg at randomisation)
2. Proteinuria (defined as greater than or equal to 0.3 g/d by 24 hour urine collection, or if a 24 hour urine collection is not available, by a urinary protein:creatinine ratio of greater than or equal to 30 mg/mmol or urinary dipstick of greater than or equal to 2+)
3. Use of an angiotensin converting enzyme (ACE) inhibitor at greater than or equal to 14+0 weeks' gestation
4. Contraindication to either arm of the trial or to pregnancy prolongation
5. Known multiple gestation
6. Known lethal or major foetal anomaly
7. Plan to terminate pregnancy
8. Prior participation in CHIPS

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 987 (Actual)
Dates: Start 2009-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Magee, MD, FRCPC, MSc, FACP, Principal Investigator — The University of British Columbia
Locations (111):
- United States (11):
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Norton Hospital Downtown, Louisville, Kentucky
  - Norton Suburban Hospital, Louisville, Kentucky
  - Beth Israel Deaconess, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Cooper University Hospital, Camden, New Jersey
  - University of North Carolina, Chapel Hill, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Meriter Hospital, Madison, Wisconsin
- Argentina (4):
  - Hospital JR Vidal, Corrientes
  - Hospital LC Lagomaggiore, Mendoza
  - Hospital Avellaneda, San Miguel de Tucumán
  - Hospital JM Cullen, Santa Fe
- Australia (6):
  - Campbelltown Hospital, Campbelltown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Women's and Children's Hospital, Adelaide
  - Ipswich Hospital, Ipswich
  - King Edward Memorial Hospital, Subiaco
  - St John of God Hospital, Subiaco
- Brazil (7):
  - Hospital Materno Infantil, Goiânia
  - Hospital Universitario Antonio Pedro, Niterói
  - Hospital Sao Lucas - PUCRS, Porto Alegre
  - Maternidade Escola da UFRJ, Rio de Janeiro
  - Clinica Perinatal Barra, Rio de Janerio
  - Laranjeiras Clinica Perinatal, Rio de Janerio
  - Maternidade Escola de Vila Nova Cachoeirinha, São Paulo
- Canada (21):
  - Calgary Health Region - Foothills Hospital, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Jim Pattison Outpatient Care and Surgery Centre, Surrey, British Columbia
  - University of British Columbia, Department of Obstetrics & Gynaecology, Vancouver, British Columbia
  - Children's & Women's Health Centre of BC, Vancouver, British Columbia
  - St Paul's Hospital, Vancouver, British Columbia
  - St Boniface General Hospital, Winnipeg, Manitoba
  - Women's Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Civic Division, Ottawa, Ontario
  - Ottawa Hospital General Division, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Hopital Sainte-Justine, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - CHUS Fleurimont, Sherbrooke, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
  - Regina General Hospital, Regina
- Chile (2):
  - Hospital Base Osorno, Osorno
  - Hospital Dr Sotero del Rio, Puente Alto
- Colombia (3):
  - Clinica Materno Infantil Farallones, Cali
  - Clinica Versalles, Cali
  - Corporacion Conmfenalco Valle - Universidad Libre, Cali
- Tartu University Hospital-Women's Clinic, Tartu, Estonia
- University of Debrecen, Debrecen, Hungary
- Israel (3):
  - Ma'ayney Hayeshua Medical Center, Bnei Brak
  - Hillel Yaffe Medical Center, Hadera
  - Nazareth Hospital (EMMS), Nazareth
- Islamic Hospital, Amman, Jordan
- Netherlands (18):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Flevo ziekenhuis, Almere Stad
  - Meander Medisch Centrum, Amersfoort
  - Academic Medical Center, Amsterdam
  - OLVG, Amsterdam
  - VU Medical Center, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - UMCG, Groningen
  - Kennemer Gasthuis Haarlem, Haarlem
  - Tergooiziekenhuizen, Hilversum
  - Spaarne Ziekenhuis, Hoofddorp
  - MUMC Maastricht, Maastricht
  - St Antonius Ziekenhuis, Nieuwegein
  - Ziekenhuis Bernhoven, Oss
  - Diakonessen Ziekenhuis, Utrecht
  - UMCU, Utrecht
  - Maxima Medical Centre, Veldhoven
  - Isala Klinieken Zwolle, Zwolle
- New Zealand (2):
  - Waitemata Health-North Shore Hospital, Auckland
  - Christchurch Women's Hospital, Christchurch
- Poland (3):
  - Medical University of Gdansk, Gdansk
  - Polish Mothers Memorial Hospital, Lodz
  - University School of Medical Sciences, Poznan
- United Kingdom (28):
  - Basildon & Thurrock University Hospital, Basildon
  - Birmingham Women's Hospital, Birmingham
  - East Lancashire Hospitals NHS Trust, Blackburn
  - Bradford Royal Infirmary, Bradford
  - Chesterfield Royal Hospital, Chesterfield
  - University Hospital Coventry and Warwickshire, Coventry
  - The Royal Derby Hospital, Derby
  - Calderdale Royal Hospital, Halifax
  - Lancashire Teaching Hospitals NHS Foundation Trust, Lancashire
  - Royal Lancaster Infirmary, Lancaster
  - Leicester Royal Infirmary, Leicester
  - Liverpool Women's Hospital, Liverpool
  - Guy's & St Thomas' Hospital, London
  - Queen Elizabeth Hospital, London
  - St Mary's Hospital, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Nottingham City Hospital, Nottingham
  - Queen's Medical Centre, Nottingham
  - King's Mill Hospital, Nottinghamshire
  - Southport & Ormskirk Hospital, Ormskirk
  - Derriford Hospital, Plymouth
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Wexham Park Hospital, Slough
  - City Hospitals Sunderland NHS Foundation Trust, Sunderland
  - Singleton Hospital, Swansea
  - South Warwickshire NHS Trust, Warwickshire
  - New Cross Hospital, Wolverhampton
  - York District Hospital, York

REFERENCES:
- [Derived] Metcalfe RK, Harrison M, Singer J, Lewisch M, Lee T, von Dadelszen P, Magee LA, Bansback N; CHIPS Study Group. Using a patient-centred composite endpoint in a secondary analysis of the Control of Hypertension in Pregnancy Study (CHIPS) Trial. Trials. 2023 Feb 7;24(1):99. doi: 10.1186/s13063-023-07118-1. PMID 36750953
- [Derived] Magee LA, Singer J, Lee T, McManus RJ, Lay-Flurrie S, Rey E, Chappell LC, Myers J, Logan AG, von Dadelszen P. Are blood pressure level and variability related to pregnancy outcome? Analysis of control of hypertension in pregnancy study data. Pregnancy Hypertens. 2020 Jan;19:87-93. doi: 10.1016/j.preghy.2019.12.002. Epub 2020 Jan 9. PMID 31927325
- [Derived] Vidler M, Magee LA, von Dadelszen P, Rey E, Ross S, Asztalos E, Murphy KE, Menzies J, Sanchez J, Singer J, Gafni A, Gruslin A, Helewa M, Hutton E, Lee SK, Lee T, Logan AG, Ganzevoort W, Welch R, Thornton JG, Moutquin JM; CHIPS Study Group. Women's views and postpartum follow-up in the CHIPS Trial (Control of Hypertension in Pregnancy Study). Eur J Obstet Gynecol Reprod Biol. 2016 Nov;206:105-113. doi: 10.1016/j.ejogrb.2016.07.509. Epub 2016 Sep 10. PMID 27665372
- [Derived] Magee LA, von Dadelszen P, Singer J, Lee T, Rey E, Ross S, Asztalos E, Murphy KE, Menzies J, Sanchez J, Gafni A, Helewa M, Hutton E, Koren G, Lee SK, Logan AG, Ganzevoort W, Welch R, Thornton JG, Moutquin JM; CHIPS Study Group*. The CHIPS Randomized Controlled Trial (Control of Hypertension in Pregnancy Study): Is Severe Hypertension Just an Elevated Blood Pressure? Hypertension. 2016 Nov;68(5):1153-1159. doi: 10.1161/HYPERTENSIONAHA.116.07862. Epub 2016 Sep 12. PMID 27620393
- [Derived] Ahmed RJ, Gafni A, Hutton EK, Hu ZJ, Pullenayegum E, von Dadelszen P, Rey E, Ross S, Asztalos E, Murphy KE, Menzies J, Sanchez JJ, Ganzevoort W, Helewa M, Lee SK, Lee T, Logan AG, Moutquin JM, Singer J, Thornton JG, Welch R, Magee LA. The Cost Implications of Less Tight Versus Tight Control of Hypertension in Pregnancy (CHIPS Trial). Hypertension. 2016 Oct;68(4):1049-55. doi: 10.1161/HYPERTENSIONAHA.116.07466. Epub 2016 Aug 22. PMID 27550914
- [Derived] Magee LA, von Dadelszen P, Rey E, Ross S, Asztalos E, Murphy KE, Menzies J, Sanchez J, Singer J, Gafni A, Gruslin A, Helewa M, Hutton E, Lee SK, Lee T, Logan AG, Ganzevoort W, Welch R, Thornton JG, Moutquin JM. Less-tight versus tight control of hypertension in pregnancy. N Engl J Med. 2015 Jan 29;372(5):407-17. doi: 10.1056/NEJMoa1404595. PMID 25629739

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 'Less Tight' Control. | 'Tight' Control.
Started | 497 | 490
Completed | 493 | 488
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 'Less Tight' Control. | 'Tight' Control. | Total
Number analyzed (Participants) | 497 | 490 | 987
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (5.7) | 33.7 (5.8) | 33.8 (5.8)
Gender [Count of Participants; unit: Participants]
  Female | 497 | 490 | 987
  Male | 0 | 0 | 0
Body-mass index [Number; unit: participants] — Available in 493 women in 'Less-tight' control, and 485 women in 'Tight' control
  participants
    <18.5 kg/m^2 | 1 | 2 | 3
    18.5-24.9 kg/m^2 | 116 | 112 | 228
    25.0-29.9 kg/m^2 | 131 | 135 | 266
    ≥30.0 kg/m^2 | 245 | 236 | 481
Cigarette smoking during this pregnancy [Number; unit: participants] | 35 | 28 | 63
Nulliparous [Number; unit: participants] — Women who were never pregnant before (i.e., first pregnancy)
  participants | 161 | 168 | 329
Weeks of gestation [Mean (Standard Deviation); unit: weeks] | 23.7 (6.3) | 24.2 (6.3) | 23.9 (6.3)
Type of nonproteinuric hypertension [Number; unit: participants]
  Preexisting hypertension | 371 | 365 | 736
  Gestational hypertension | 126 | 125 | 251
Prior blood pressure ≥160 mm Hg systolic or ≥110 mm Hg diastolic during this pregnancy [Number; unit: participants] | 82 | 59 | 141
Antihypertensive medication at enrollment [Number; unit: participants] | 279 | 287 | 566
Blood pressure within 1 wk before randomization [Mean (Standard Deviation); unit: mmHg]
  Systolic | 140.4 (9.7) | 139.7 (9.8) | 140.1 (9.8)
  Diastolic | 92.6 (4.8) | 92.2 (5.2) | 92.4 (5.0)
Currently monitoring blood pressure at home [Number; unit: participants] | 185 | 194 | 379
Gestational diabetes at enrollment [Number; unit: participants] | 32 | 31 | 63

OUTCOME MEASURES:

1. Primary Outcome: Pregnancy Loss or NICU Admission for Greater Than 48 Hours
Description: Pregnancy loss or NICU admission for greater than 48 hours, as recorded in the maternal and infant medical records immediately following the birth (or pregnancy loss), and then again after the mothers' and infants' discharge home. Supplemental information, about potential post-discharge maternal or neonatal morbidities in the 6 weeks following birth for the mother, or 28 days of life for the baby, will be obtained by contacting women at 6 weeks postpartum and/or from medical records.
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | 'Less Tight' Control. | 'Tight' Control.
Number analyzed (Participants) | 493 | 488
participants | 155 | 150
Statistical Analysis 1: Comparison: 'Less Tight' Control. vs 'Tight' Control; We estimated that with a sample size of 514 per group, the study would have 80% power, at a two-tailed alpha level of 0.05, assuming primary outcome rates of 33% in the tight-control group and 25% in the less-tight-control group, a 10% rate of crossover, a 1% loss to follow-up, and two interim analyses, as calculated with the chi-square test with the use of East software (Cytel) and the Lan-DeMets spending function with O'Brien-Fleming-type boundaries for early stopping; Test type: Superiority or Other; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.77 to 1.35]

2. Secondary Outcome: Serious Maternal Complications Measured up to 6 Weeks Postpartum
Description: Serious maternal complications measured up to 6 weeks postpartum. Death or one or more life-threatening maternal complications:
  1. Adverse neurological complications (stroke, eclampsia, and/or blindness), and/or
  2. End-organ failure (uncontrolled hypertension, inotropic support, pulmonary oedema, respiratory failure, myocardial ischaemia/infarction, renal failure, coagulopathy, and/or transfusion)
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | 'Less Tight' Control. | 'Tight' Control.
Number analyzed (Participants) | 493 | 488
participants | 18 | 10
Statistical Analysis 1: Comparison: 'Less Tight' Control. vs 'Tight' Control; Test type: Superiority or Other; Odds Ratio (OR) = 1.74, 95% CI 2-sided [0.79 to 3.84]

ADVERSE EVENTS:
Arm/Group | 'Less Tight' Control. | 'Tight' Control.
Serious Adverse Events (participants affected / at risk) | 155/493 | 150/488
Other Adverse Events (participants affected / at risk) | 241/493 | 223/488
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 'Less Tight' Control. (N=493) | 'Tight' Control. (N=488)
Pregnancy loss (Pregnancy, puerperium and perinatal conditions) | 15 | 15
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0
Elective termination (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Perinatal death (Pregnancy, puerperium and perinatal conditions) | 14 | 11
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 12 | 7
Neonatal death (Pregnancy, puerperium and perinatal conditions) | 2 | 4
High-level neonatal care for >48hr (Pregnancy, puerperium and perinatal conditions) | 141/480 | 139/479
Birthweight <10th percentile (Pregnancy, puerperium and perinatal conditions) | 79/491 | 96
Birthweight <3rd percentile (Pregnancy, puerperium and perinatal conditions) | 23/491 | 26
Uncontrolled hypertension (Cardiac disorders) | 0 | 0
Transient ischemic attack or stroke (Nervous system disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Transfusion (Blood and lymphatic system disorders) | 16 | 8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 'Less Tight' Control. (N=493) | 'Tight' Control. (N=488)
Placental abruption (Pregnancy, puerperium and perinatal conditions) | 11 | 11
Severe hypertension (Cardiac disorders) | 200 | 134
Preeclampsia (Pregnancy, puerperium and perinatal conditions) | 241 | 223

LIMITATIONS AND CAVEATS:
Women with preexisting or gestational hypertension included, and may have differing management. Primary/secondary outcomes included causes of pregnancy loss and interventions for neonatal care not expected to be associated with maternal BP control

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No